CLINICAL TRIAL: NCT05291455
Title: Efficacy of Lacosamide in Neonatal Status Epilepticus: A Randomized Controlled Study
Brief Title: Lacosamide in Neonatal Status Epilepticus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, ass prof tropical medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: abeer ped neurology
Record Dates: First submitted 2022-03-18; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide; Phenobarbital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lacosamide (Experimental): Lacosamide will be given.
  Interventions: Drug: Lacosamide
- Phenobarbitone (Active Comparator): Phenobarbital will be given
  Interventions: Drug: Phenobarbital

INTERVENTIONS:
Drug: Lacosamide — lacosamide will be given
  Other Names: lacosa
  Arms: Lacosamide
Drug: Phenobarbital — phenobarbital will be given
  Other Names: phenobarbitone
  Arms: Phenobarbitone

SUMMARY:
Lacosamide in neonatal status epilepticus

DETAILED DESCRIPTION:
The study will assess the efficacy of Lacosamide in neonatal status epilepticus

ELIGIBILITY:
Inclusion Criteria:

* neonates with status epilepticus

Exclusion Criteria:

* congenital anomalies or organ dysfunction

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
number of children with cessation or improved duration of status epilepticus | 1 year
  the number of children with cessation or improved duration of status epilepticus

CONTACTS AND LOCATIONS:
Overall Officials: abeer salamah, lecturer, Principal Investigator — Kafrelsheikh University
Locations (1):
- Kafrelsheikh University, Tanta, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No